CLINICAL TRIAL: NCT06580444
Title: Brexanolone to Target Concurrent Posttraumatic Stress Disorder (PTSD) and Stress Induced Alcohol Use in Veterans: A Dose Finding Study
Brief Title: Brexanolone to Target Concurrent PTSD and Stress Induced Alcohol Use in Veterans: A Dose Finding Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacotherapies for Alcohol and Substance Use Disorders Alliance (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Congressionally Directed Medical Research Programs (U.S. Federal Agency); VA Connecticut Healthcare System (U.S. Federal Agency); Sage Therapeutics (Industry); RTI International (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AS210006-A09
Record Dates: First submitted 2024-07-25; First posted 2024-08-30 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use Disorder (AUD); Post Traumatic Stress Disorder (PTSD)
Keywords: Alcohol Used Disorder (AUD); Post Traumatic Stress Disorder (PTSD); Alcohol Use; Heavy Drinkers; Brexanolone
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic; Alcohol Drinking | interventions — brexanolone

STUDY DESIGN:
Intervention Model Description: At baseline, participants who meet eligibility criteria are randomized to placebo or 90, 60, or 30 mcg/kg/h doses of BREX along with the order/sequence of their stress and neutral lab sessions in a double-mask fashion for the duration of the study. The treatment allocation will be equal in each arm. Additionally, the order/sequence of stress and neutral laboratory sessions will be randomized for laboratory sessions (e.g., if stress on session #1 then neutral on session #2) in a manner that assures treatment balance within laboratory session.
  Each participant will be randomized to receive a target dose of either 90, 60, 30 and 0 mcg/kg/h, titrated over the 20 hours; both the 90 and 60 doses have shown efficacy to target postpartum depressive symptoms and the 30 mcg/kg/h will test the lower limits of efficacy.
  The sample size will have 10 participants in each group for doses 0, 30, 60 and 90 to equal 40 participants.
Who Masked: Participant, Care Provider, Investigator
Masking Description: To minimize bias, a placebo drug is employed as the comparison group to active study drug doses and the study is conducted in a double-masked fashion in that both the participants and anyone assessing study outcomes are masked to treatment assignment. The only individuals at the site with access to treatment assignment information are the research pharmacists.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (No Intervention): A 0.9% bag of sodium chloride will be administered intravenously. Participant will be given a self-administered alcoholic drink of their choice that is individually calculated, and they will receive money up to $15 for every minute they resist drinking.
- 90mcg/kg/h dose of Brexanolone (Active Comparator): Brexanolone will be diluted with sterile water and 0.9% sodium chloride and will be administered intravenously. Participant will be given a self-administered alcoholic drink of their choice that is individually calculated, and they will receive money up to $15 for every minute they resist drinking.
  Interventions: Drug: Brexanolone
- 60mcg/kg/h dose of Brexanolone (Active Comparator): Brexanolone will be diluted with sterile water and 0.9% sodium chloride and will be administered intravenously. Participant will be given a self-administered alcoholic drink of their choice that is individually calculated, and they will receive money up to $15 for every minute they resist drinking.
  Interventions: Drug: Brexanolone
- 30mcg/kg/h dose of Brexanolone (Active Comparator): Brexanolone will be diluted with sterile water and 0.9% sodium chloride and will be administered intravenously. Participant will be given a self-administered alcoholic drink of their choice that is individually calculated, and they will receive money up to $15 for every minute they resist drinking.
  Interventions: Drug: Brexanolone

INTERVENTIONS:
Drug: Brexanolone — The participant will receive either a placebo, or 90, 60, or 30 mcg/kg/hr of Brexanolone over a 20-hour period intravenous infusion.
  Other Names: Placebo
  Arms: 30mcg/kg/h dose of Brexanolone; 60mcg/kg/h dose of Brexanolone; 90mcg/kg/h dose of Brexanolone

SUMMARY:
The purpose of this research study is to find out how Zulresso®/brexanolone influences Posttraumatic Stress Disorder (PTSD) symptoms and alcohol use.

DETAILED DESCRIPTION:
The overall objectives of this study are to establish the safety of administering 90, 60, and 30mcg/kg/h target doses of brexanolone (BREX; 20-hour infusion; versus placebo) and investigate efficacy of each dose to reduce PTSD symptoms, alcohol consumption, and stress reactivity via mood-induction paradigms in individuals with PTSD/AUD.

The primary aims of this study are to:

1. Evaluate the safety and tolerability of BREX 90, 60, and 30 mcg/kg/h among individuals with PTSD/AUD
2. Investigate the medication effect of the 90, 60, and 30 mcg/kg/h doses of BREX to reduce alcohol consumption and PTSD symptoms in men and women with PTSD/AUD.

The secondary aim of this study is to:

1. Investigate the medication effect of each of the 90, 60, 30 mcg/kg/h doses of BREX to reduce stress reactivity via mood-induction paradigm in men and women with PTSD/AUD.

The exploratory aim of this study is to:

1. Explore sex-specific responses to brexanolone's effect on PTSD and alcohol use among men and women with PTSD/AUD.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 21-70 years old, either active duty or with a history of US military service.
4. Current DSM-5 diagnostic criteria for AUD (mild, moderate, or severe) within 6 months at the time of the intake, as measured via Quick Structured Clinical Interview for DSM-5 (QuickSCID-5), as well as the following drinking criteria (measured by the Timeline Followback):

   1. Men: drink greater than 14 drinks per week and exceed five drinks per day at least once per week within the past 30 days at the time of intake.
   2. Women: drink greater than 7 drinks per week and exceed four drinks per day at least once per week within the past 30 days at the time of intake.
   3. Men and women will not endorse a desire to completely abstain from alcohol use at any point during the study. It will be necessary to confirm, via self-report (TLFB), consumption of alcohol within the week prior to the alcohol laboratory sessions. In the event the TLFB indicates recent abstinence, participants will be explicitly queried regarding desire to completely abstain from alcohol use moving forward, utilizing a one question item. If a patient completes the drug administration session, but then endorses desire to abstain completely he/she will be followed via observation and not participate in laboratory sessions, in which alcohol is self-administered.
5. Have a Clinician Administered PTSD Scale for DSM-5 (CAPS-5) total score ≥26 for the past month at intake, as well as a PTSD Checklist for DSM-5 (PCL-5) total score ≥31 for the past month at intake.
6. Not currently taking medications thought to influence alcohol consumption such as Acamprosate, formulations of naltrexone, topiramate, ondansetron, baclofen, disulfiram, or gabapentin within 30 days prior to enrollment.
7. Females of childbearing potential, who are not surgically sterilized (tubal ligation/hysterectomy) or not post-menopausal (no menstrual period for > 6 months) must be willing to use a medically acceptable and effective birth control method for at least 1 month prior to screening, randomization and intake and while participating in the study. Medically acceptable methods of contraception that may be used by the participant include abstinence, birth control pills, patches, implants, injections, rings, diaphragm, intrauterine device (IUD), or condoms.

Exclusion Criteria:

1. Meets current DSM-5 diagnostic criteria for schizophrenia, bipolar disorder, and/or other severe mental illnesses, as defined by the QuickSCID-5 at intake. Please note that the QuickSCID-5 provides a Psychotic Symptom Screen. In the event, a patient screens positive for psychotic symptoms, the study team member will administer Modules B (Psychotic and Associated Symptoms) and C (Differential Diagnosis of Psychotic Disorders) from the Structured Clinician Interview for DSM-5 Clinician Version to determine a diagnosis of schizophrenia or another psychotic disorder.
2. Increased risk of suicide that necessitates inpatient treatment or warrants therapy excluded by the protocol, and/or a current suicidal plan, per investigator's clinical judgement during interview.
3. Treatment with trauma-focused therapy (e.g., Cognitive Processing Therapy, Prolonged Exposure Therapy, or Eye Movement Desensitization & Reprocessing Therapy) for PTSD within two weeks of intake (if participant is receiving therapy, he/she must complete treatment prior to entering study). Note: Supportive psychotherapy in process at time of Screening may be continued.
4. Meets criteria for current diagnosis of moderate or severe non-alcohol substance use disorder (except for caffeine and nicotine), as measured via QuickSCID-5, during the preceding 1 month relative to intake, per PI discretion, based on participant's screening interview.
5. Tests positive for illicit substances during urine toxicology screens (except cannabis) at intake session. Patients who utilize cannabis but do not meet substance use disorder criteria are permitted.
6. Self-reported past 30-day use at intake of psychoactive drugs (except cannabis), including opioids, CNS depressants (such as benzodiazepines), use of psychotropic medications in the class of antipsychotics, mood stabilizers, or stimulants. Note: Participant use of stable doses (prescribed for >2 months and the current dose has been stable or ≥3 weeks at intake) of antidepressants will be reviewed by Study MD.
7. Likely to exhibit clinically significant alcohol withdrawal during the study. Specifically, we will exclude subjects who a) have a history of perceptual distortions, seizures, delirium, or hallucinations upon withdrawal, assessed during physical examination as part of intake procedures or b) have a score of > 8 on the Clinical Institute Withdrawal Assessment scale at intake appointment. Participants must have a CIWA-Ar score of < 8 prior to randomization.
8. Any clinically significant, uncontrolled, or medical/surgical condition, that at the discretion of the investigator, would contraindicate use of brexanolone, or limit ability to complete study assessments, including end stage renal disease, significant arrhythmia or heart block, or heart failure, severe thrombocytopenia or hemophilia, severe hepatic failure, complete hearing loss, and/or need for surgery that might interfere with ability to participate. Such conditions will be assessed by the Study MD based upon physical examination (including review of medical history), as well as review of medical records, ECG and basic blood chemistries (i.e., CBC).
9. Females who are pregnant, nursing, planning to become pregnant or fail to use one of the following methods of birth control during study participation (unless she or her partner is surgically sterile, or she is postmenopausal). Birth control includes: hormonal contraceptives (oral, implant, injection, patch, or ring), contraceptive sponge, double barrier (diaphragm or condom plus spermicide) or IUD.
10. Any finding that, in the view of the principal investigator, would compromise the subject's ability to fulfill the study visit schedule or requirements.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-28 (Estimated); Primary Completion 2027-02-26 (Estimated); Study Completion 2027-03-19 (Estimated)

PRIMARY OUTCOMES:
Severity and numbers of treatment-emergent AEs | From onset of Brexanolone administration until 30-day follow up.
  The number and proportion of individuals experiencing any adverse event, any SAE, and any related adverse event overall will be summarized using frequency tables. No formal statistical tests will be conducted, rather the safety will be evaluated from a risk/benefit perspective. Any p-values reported will be for descriptive purposes only.
Change in Heart Rate from onset of Brexanolone administration until discharge from the drug administration session. | An average of 22 hours (From the start of Brexanolone administration on day 1 at 10 am until 7 am on day 2)
  The change in heart rate a physiological safety/stress measure are continuous and obtained multiple times after study drug administration which occurs on day 1. This measure will be analyzed using descriptive statistics and graphical summaries including time-specific summary statistics (e.g., box and whisker plots).
Change in Blood Pressure from onset of Brexanolone administration until discharge from the drug administration session. | An average of 22 hours (From the start of Brexanolone administration on day 1 at 10 am until 7 am on day 2)
  The change in blood pressure a physiological safety/stress measure are continuous and obtained multiple times after study drug administration which occurs on day 2. This measure will be analyzed using descriptive statistics and graphical summaries including time-specific summary statistics (e.g., box and whisker plots).
Change in Cortisol from onset of Brexanolone administration until discharge from the drug administration session. | FAn average of 22 hours (From the start of Brexanolone administration on day 1 at 10 am until 7 am on day 2)
  The change in Cortisol a physiological safety/stress measure are continuous and obtained multiple times after study drug administration which occurs on day 2. This measure will be analyzed using descriptive statistics and graphical summaries including time-specific summary statistics (e.g., box and whisker plots).
Change in percentage of milliliters of alcohol consumed during the 2-hour ad-libitum drinking paradigm between laboratory sessions (stress vs. neutral). | During the 2-hour ad-libitum drinking paradigm between lab sessions (stress Vs Neutral)
  A set of dose-response models will be tested response using the Multiple Comparisons Procedure Modifications (MCP-Mod) methodology including change in percentage of milliliters consumed during the 2-hour ad-libitum drinking paradigm within laboratory sessions (stress and neutral) as dependent variable, the treatment as factor (90, 60, 30 and 0 mcg/kg/h), and baseline dependent value. These dose-response models with repeated measures will be used to test the effects of the regimens of 90, 60, and 30 mcg/kg/h doses of brexanolone on alcohol consumption in self-administration.
Change in Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) score from intake until 30-day follow-up | From intake, day 0 through day 37 (30-day follow-up).
  Another set of dose-response models will test Multiple Comparisons Procedure Modifications (MCP-Mod) methodology for the 30-day follow-up in PCL-5 score as dependent variable, the treatment as factor (90, 60, 30 and 0 mcg/kg/h), and baseline dependent value. These dose-response models will be used to test the effects of the regimens of 90, 60, 30 and 0 mcg/kg/h doses of brexanolone on PTSD symptoms.
  Scale PCL-5 is 0-4 with 0 being not at all and 4 being extreme; the higher score is worse outcome
Change in Change in Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) score from intake until end of dosing. | An average of 22 hours (From intake, day 0 through end of infusion on Day 2)
  Another set of dose-response models will test Multiple Comparisons Procedure Modifications (MCP-Mod) methodology including change from intake to end of dosing in PCL-5 score as dependent variable, the treatment as factor (90, 60, 30 and 0 mcg/kg/h), and baseline dependent value. The same modeling will be repeated for the 30-day follow-up timepoint. These dose-response models will be used to test the effects of the regimens of 90, 60, 30 and 0 mcg/kg/h doses of brexanolone on PTSD symptoms.
  Scale PCL-5 is 0-4 with 0 being not at all and 4 being extreme; the higher score is worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: MacKenzie R. Peltier, Ph.D., Principal Investigator — Assistant Professor Psychiatry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PASA Website — http://pasa-research.org/